CLINICAL TRIAL: NCT04547348
Title: Efficacy of Treatment With DENOsumab of an Acute CHARCOT Foot in Patients With Diabetes. A Multicenter, Double-blind, Randomized, Placebo-controlled Trial.
Brief Title: The DENOCHARCOT Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ole Lander Svendsen (Other)
Responsible Party: Sponsor-Investigator, Ole Lander Svendsen, Professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CODIF-008
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Charcot Foot; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab treated group (Experimental): Participants will receive a 60 mg subcutaneous injection of Prolia upon randomization and on week 28 after the first injection provided remission of the Charcot foot has not been achieved by then
  Interventions: Drug: Denosumab Injection
- Placebo treated group (Placebo Comparator): Participants will receive an injection of placebo (saline) instead of Prolia
  Interventions: Drug: Denosumab Injection

INTERVENTIONS:
Drug: Denosumab Injection — Injections made subcutaneously per standard description

SUMMARY:
The aim of the present trial is to assess the efficacy of treatment of acute Charcot foot in diabetes patients with Prolia® on clinical relevant Outcomes in a randomized, double blind, placebo-controlled trial.

DETAILED DESCRIPTION:
After giving informed consent and being enrolled, patients will be randomized to one of two group given either Denosumab treatment or injection with placebo. The patients will then undergo a 52 week follow up with regular controls to asses if clinical signs of Charcot is in remission, which will be verified using relevant radiological modalities. Upon final visit the patients will be examined using radiology, blood samples, biothesiometry and objective examinations, following up on the same examinations being made upon inclusion.

Primary outcome will be time until full remission of the Charcot foot defined as clinical healing (The acute Charcot foot is clinically healed when the temperature difference at the site maximum temperature on the affected Charcot foot is < 2 degrees Celsius compared to the similar site on the contra-lateral foot, measured using an infrared thermometer, and edema and redness of the skin has subsided) followed up by radiological signs of healing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Type 1 or type 2 diabetes (diagnosed diabetes for more than 3 months)
* Diagnosed with acute Charcot foot defined as a unilateral red, swollen and warm foot, with a difference of skin temperature of more than 2 °C compared with the unaffected foot and with sign of Charcot on either x-rays of the foot, MRI, bone scintigram or PET/CT.
* Peripheral neuropathy: Previously diagnosed and/or biothesiometri: > 25 V or lack of sensation of 10 grams monofilament on 1. toe at the acute Charcot foot.

Exclusion Criteria:

* Duration of the acute Charcot foot for more than 3 months (at the screening visit).
* Existing foot ulcer on the affected foot
* Previous acute or chronic Charcot of the affected foot
* Planned surgery on the acute Charcot foot
* Infection (cellulitis or osteomyelitis) of the affected foot (clinically and/or radiologically proven)
* Previous midfoot or proximal to mid foot amputation of the affected foot
* Hypocalcemia (Serum Calcium <2.1 mmol/L or Calcium ion < 1.12 mmol/L)
* Vitamin D deficiency (Serum 25-hydroxyvitamin D < 50 nmol/L)
* Renal failure (serum creatinine >200 mmol/L or eGFR < 30 ml/min).
* Treatment with Denosumab within the last 12 months. • Have a known hypersensitivity to Denosumab • History of osteonecrosis of the jaw.
* Poor oral hygiene, which is defined as within 3 months of a tooth extraction, dental implants or mandibular surgery
* Planned mandibular surgery or dental implants within the next 12 months.
* Prior non-traumatic vertebral fracture
* Treatment with medication known to affect bones within the last 12 months (such as bisphosphonates, Forsteo®, calcitonin, Protelos®, selective estrogen receptor modulators, glucocorticoids and sex hormones)
* Active or chronic liver disease *Chronic liver disease is defined as clinical history of decompensated chronic liver disease (ascites, encephalopathy or variceal bleeding) *Acute Liver disease is defined as an INR of > 1.5 (in the absence of the use of Warfarin) and AST and ALT > 2 x ULN
* History of inflammatory arthropathies (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, autoimmune arthropathy)
* Pre-existing medical condition judged to preclude safe participation in the study
* Current treatment with cytotoxic drugs or with systemically administered glucocorticoids
* Abuse of alcohol or drugs, or presence of any condition that in the Investigators opinion may lead to poor adherence to study protocol
* Pregnancy, breast feeding or planning pregnancy or not using adequate contraceptive methods. The following contraceptive products are considered to be safe: Intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long-acting injections).
* Likely inability to comply with the visits because of planned activity
* Use of any investigational product with the last month.
* Use of any drug or any other reason which in the Investigator's opinion could interfere with the outcome of the treatment of the acute Charcot foot.
* Cancer, or any clinically significant disease or disorder, except for conditions associated to the diabetes, which in the Investigator's opinion could interfere with the results of the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Time until remission | 52 weeks
  Time from first injection of IP until the time point where the acute Charcot foot is clinically healed/in remission, ie. the temperature difference at the site maximum temperature on the affected Charcot foot is < 2 degrees Celsius compared to the similar site on the contra-lateral foot, measured using an infrared thermometer, and edema and redness of the skin has subsided - at two subsequent visits 4 weeks apart. The off-loading regime will be continued until the second visit. The first of the two visits is the timepoint of healing of the acute Charcot foot.

SECONDARY OUTCOMES:
Fraction of clinical healed participants at each study visit. | 52 weeks
Fraction of healing on X-rays and MRI (or PET/CT or Scintigram) at the time of clinical healing and at the End of trial. | 52 weeks
Number of relapses (defined as need for/prescription of off- loading with cast of the Charcot foot again) | 52 weeks
Time without relapse (the time from clinical healing/remission to the relapse or to End of Trial at 12 months). | 52 weeks
Number of patients with development of complications to the acute Charcot foot, as well as number of development of foot ulcer, deformity, need for special footwear or surgery and fractures of bones in the foot, respectively. | 52 weeks
Changes in BMD (lumbar spine, hip) | 52 weeks
Changes in markers of bone turnover (CTX and P1NP) | 52 weeks
Changes in markers of glycemic control (HbA1c) | 52 weeks
Incidence of Adverse Events and Serious Adverse Events | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ole Lander Svendsen, MD, Study Chair — Region Hovedstadens Apotek
Locations (8):
- Denmark (8):
  - Steno Diabetes Center North, Aalborg
  - Steno Diabetes Center Aarhus, Aarhus
  - Bispebjerg Hospital, Copenhagen NV
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Nordsjællands Hospital, Hillerød
  - Hvidovre hospital, Hvidovre
  - Zealand University Hospital, Køge
  - Steno Diabetes Center Odense, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeffcoate WJ. Charcot foot syndrome. Diabet Med. 2015 Jun;32(6):760-70. doi: 10.1111/dme.12754. Epub 2015 Apr 15. PMID 25818542
- [Background] Christensen TM, Gade-Rasmussen B, Pedersen LW, Hommel E, Holstein PE, Svendsen OL. Duration of off-loading and recurrence rate in Charcot osteo-arthropathy treated with less restrictive regimen with removable walker. J Diabetes Complications. 2012 Sep-Oct;26(5):430-4. doi: 10.1016/j.jdiacomp.2012.05.006. Epub 2012 Jun 12. PMID 22699112
- [Background] Pitocco D, Ruotolo V, Caputo S, Mancini L, Collina CM, Manto A, Caradonna P, Ghirlanda G. Six-month treatment with alendronate in acute Charcot neuroarthropathy: a randomized controlled trial. Diabetes Care. 2005 May;28(5):1214-5. doi: 10.2337/diacare.28.5.1214. No abstract available. PMID 15855594
- [Background] Anderson JJ, Woelffer KE, Holtzman JJ, Jacobs AM. Bisphosphonates for the treatment of Charcot neuroarthropathy. J Foot Ankle Surg. 2004 Sep-Oct;43(5):285-9. doi: 10.1053/j.jfas.2004.07.005. PMID 15480402
- [Background] Jude EB, Selby PL, Burgess J, Lilleystone P, Mawer EB, Page SR, Donohoe M, Foster AV, Edmonds ME, Boulton AJ. Bisphosphonates in the treatment of Charcot neuroarthropathy: a double-blind randomised controlled trial. Diabetologia. 2001 Nov;44(11):2032-7. doi: 10.1007/s001250100008. PMID 11719835
- [Background] Bem R, Jirkovska A, Fejfarova V, Skibova J, Jude EB. Intranasal calcitonin in the treatment of acute Charcot neuroosteoarthropathy: a randomized controlled trial. Diabetes Care. 2006 Jun;29(6):1392-4. doi: 10.2337/dc06-0376. No abstract available. PMID 16732029
- [Background] Pakarinen TK, Laine HJ, Maenpaa H, Mattila P, Lahtela J. The effect of zoledronic acid on the clinical resolution of Charcot neuroarthropathy: a pilot randomized controlled trial. Diabetes Care. 2011 Jul;34(7):1514-6. doi: 10.2337/dc11-0396. Epub 2011 May 18. PMID 21593295
- [Background] Petrova NL, Dew TK, Musto RL, Sherwood RA, Bates M, Moniz CF, Edmonds ME. Inflammatory and bone turnover markers in a cross-sectional and prospective study of acute Charcot osteoarthropathy. Diabet Med. 2015 Feb;32(2):267-73. doi: 10.1111/dme.12590. Epub 2014 Oct 17. PMID 25251588
- [Background] Jansen RB, Christensen TM, Bulow J, Rordam L, Jorgensen NR, Svendsen OL. Markers of Local Inflammation and Bone Resorption in the Acute Diabetic Charcot Foot. J Diabetes Res. 2018 Aug 2;2018:5647981. doi: 10.1155/2018/5647981. eCollection 2018. PMID 30155488
- [Background] Busch-Westbroek TE, Delpeut K, Balm R, Bus SA, Schepers T, Peters EJ, Smithuis FF, Maas M, Nieuwdorp M. Effect of Single Dose of RANKL Antibody Treatment on Acute Charcot Neuro-osteoarthropathy of the Foot. Diabetes Care. 2018 Mar;41(3):e21-e22. doi: 10.2337/dc17-1517. Epub 2017 Dec 22. No abstract available. PMID 29273577
- [Background] Tsourdi E, Langdahl B, Cohen-Solal M, Aubry-Rozier B, Eriksen EF, Guanabens N, Obermayer-Pietsch B, Ralston SH, Eastell R, Zillikens MC. Discontinuation of Denosumab therapy for osteoporosis: A systematic review and position statement by ECTS. Bone. 2017 Dec;105:11-17. doi: 10.1016/j.bone.2017.08.003. Epub 2017 Aug 5. PMID 28789921
- See also: Prolia product summary — https://www.ema.europa.eu/en/documents/product-information/prolia-epar-product-information_en.pdf
- See also: Xgeva product summary — https://www.ema.europa.eu/en/medicines/human/EPAR/xgeva